CLINICAL TRIAL: NCT01110863
Title: Characterization of Proliferating Compartment in B-Cell Patients and in Healthy Aging Subjects
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Nicholas Chiorazzi, Investigator, The Feinstein Institute for Medical Research, Northwell Health
Other Study IDs: 05-05-096; GAC # 0117 (Other: GAC # 0117)
Record Dates: First submitted 2009-12-10; First posted 2010-04-27 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood cells, Bone Marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Lymphocytic Leukemia: Chronic Lymphocytic Leukemia

SUMMARY:
By ingesting a non-radioactive and non-toxic compound "heavy water" for 6 weeks, the DNA of newly developed cells in the body of subjects with B-cell chronic lymphocytic leukemia can be labeled and followed by performing routine blood draws at specified time intervals. By using mass spectrometric analysis we can measure how quickly new B-CLL cells are generated in the bone marrow and how quickly they leave the blood, a measure of cell turnover. This will help us to better understand the unique characteristics of this disease process.

DETAILED DESCRIPTION:
By ingesting a non-radioactive and non-toxic compound "heavy water" for 6 weeks, the DNA of newly developed cells in the body of subjects with B-cell chronic lymphocytic leukemia (B-CLL) can be labeled and followed by performing routine blood draws at specified time intervals. By using mass spectrometric analysis we can measure how quickly new B-CLL cells are generated in the bone marrow and how quickly they leave the blood, a measure of cell turnover. This will help us to better understand the unique characteristics of this disease process.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age,
* Patients must be willing to contribute the required amount of blood without compromising their well being,
* Participants must be willing to be contacted in the future.

Exclusion Criteria:

* Pregnancy,
* Patients who are known to be anemic, with a hemoglobin < 8,
* Patients who are known to be infected with HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic Lymphocytic Luekemia
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2005-12; Primary Completion 2016-02-12 (Actual); Study Completion 2016-02-12 (Actual)

PRIMARY OUTCOMES:
Characterization of the Proliferating Compartment in B-CLL Patients and in Healthy Aging Subjects | 1 year
  B-CLL is a dx of accumulation rather than proliferation. Evidence for various forms of clonal evolution suggests that B-CLL clones may be more dynamic than previously assumed. A non-radioactive, stable isotopic labeling method to measure B-CLL cell kinetics in vivo. Subjects drank an aliquot of 2H2O daily for 84 days, and 2H incorporation into the deoxyribose moiety of DNA of their newly divided B-CLL cells, measured by gc/ms, during the labeling period. Birth rates were calculated from the kinetic profiles. Death rates were defined as the difference between calculated birth and growth rates.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Chiorazzi, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States